CLINICAL TRIAL: NCT04245085
Title: A Randomised Non-comparative Open Label Phase II Trial of Atezolizumab Plus Bevacizumab, With Carboplatin-paclitaxel or Pemetrexed, in EGFR-mutant Non-small Cell Lung Carcinoma With Acquired Resistance
Brief Title: ABC-lung: Atezolizumab, Bevacizumab and Chemotherapy in EGFR-mutant Non-small Cell Lung Carcinoma
Acronym: ABC-lung
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ETOP IBCSG Partners Foundation (Network)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ETOP 15-19; MO40586 (Other: F. Hoffmann-La Roche Ltd. Number)
Record Dates: First submitted 2019-12-16; First posted 2020-01-28 (Actual); Last update posted 2025-01-08 (Actual); Status verified 2025-01

CONDITIONS: EGFRmutant Stage IIIB/C or IV Non-squamous NSCLC
MeSH Terms: interventions — atezolizumab; Bevacizumab; Carboplatin; Paclitaxel; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Active Comparator): * Atezolizumab (1200 mg) Q3W, until PD
  * Bevacizumab (15 mg/kg), Q3W, until PD
  * Carboplatin (AUC5) Q3W, 4-6 cycles
  * Paclitaxel (175-200 mg/m2), Q3W, 4-6 cycles
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Carboplatin; Drug: Paclitaxel
- Arm B (Active Comparator): * Atezolizumab (1200 mg), Q3W, until PD
  * Bevacizumab (15 mg/kg), Q3W, until PD
  * Pemetrexed (500 mg/m2), Q3W, until PD
  Interventions: Drug: Atezolizumab; Drug: Bevacizumab; Drug: Pemetrexed

INTERVENTIONS:
Drug: Atezolizumab — Patients in both treatment arms will receive atezolizumab at a fixed dose of 1200 mg i.v. on day one of every 3-week (3 days) cycle, until progression of disease determined according to RECIST v1.1 or lack of tolerability, or patient declines further treatment.
  Treatment beyond RECIST-defined progression will be allowed if patient is continuing to derive clinical benefit.
  Other Names: Tecentriq
Drug: Bevacizumab — Patients in both treatment arms will receive bevacizumab at a dose of 15 mg/kg i.v. on day one of every 3-week (+/- 3 days) cycle, until progression of disease determined according to RECIST v1.1 or lack of tolerability, or patient declines further treatment.
  Other Names: Avastin
Drug: Carboplatin — Patients in treatment Arm A will receive carboplatin, AUC5 every 3 weeks for 4-6 cycles.
  Arms: Arm A
Drug: Paclitaxel — Patients in treatment Arm A will receive paclitaxel, 175-200 mg/m2 (at the investigators' discretion), every 3 weeks for 4-6 cycles.
  Arms: Arm A
Drug: Pemetrexed — Patients in treatment Arm B will receive Pemetrexed, 500 mg/m2 every 3 weeks until progression of disease determined according to RECIST v1.1 or lack of tolerability, or patient declines further treatment.
  Other Names: Alimta
  Arms: Arm B

SUMMARY:
ETOP 15-19 ABC-lung is an international, multi-centre open-label, randomized phase II trial with two non-comparative parallel arms of atezolizumab plus bevacizumab with carboplatin-paclitaxel (Arm A) or atezolizumab, bevacizumab and pemetrexed (Arm B) in patients with stage IIIB-IV non-squamous non-small cell lung cancer (NSCLC) harbouring EGFR mutations after failure of standard EGFR tyrosine kinase inhibitors (TKIs).

ELIGIBILITY:
Inclusion Criteria:

1. Patients (male/female) must be ≥18 years of age.
2. Chemotherapy naïve, non-squamous NSCLC, stage IIIB/C (not amenable to radical therapy) or IV. Patients who have received previous adjuvant or neoadjuvant chemotherapy are eligible if the date of last dose of treatment was at least 12 months before randomisation.
3. Known EGFR mutations genotypes by tissue or ctDNA, patients with common mutations (L858R or Del19) and other rare mutations (e.g. S768I, G719X) are eligible.
4. Measurable or evaluable disease by RECIST v1.1.
5. Disease progression (during or after) or unacceptable side effects from prior treatment with at least one EGFR TKI (washout period = 7 days).

   If most recent line of treatment (1st or 2nd line) was a third-generation EGFR TKI (e.g. osimertinib):
   * Patient must be known to be EGFR mutation positive, either on fresh tumour biopsy taken >7 days prior to protocol treatment start or by recent ctDNA analysis (informative ctDNA test, local test).
   * T790M genotype is allowed

   If most recent line of treatment (1st or 2nd line) was a first- or second-generation EGFR TKI (e.g. afatinib, dacomitinib, erlotinib, gefitinib):

   - Patient must be known to be tissue EGFR T790M wild type (local test) on most recent line of EGFR TKI or if no tissue re-biopsy, no evidence of T790M on ctDNA but identified L858R, del19, S768I or G719X genotypes (informative ctDNA test, local test)
6. Treatment with an EGFR TKI therapy for at least 30 days
7. Adequate haematological function:

   * Haemoglobin greater or equal 90 g/L
   * Absolute neutrophils count (ANC) greater or equal 1.5× 109/L
   * Platelet count greater or equal 100× 109/L
8. Adequate renal function:

   • Creatinine clearance greater or equal 45 mL/min (using the Cockcroft-Gault formula)
9. Adequate liver function:

   * ALT and AST less or equal 2.5× ULN. If the patient has liver metastases, ALT and AST must be less or equal 5× ULN
   * Total bilirubin less or equal 1.5x ULN.
10. Willingness to provide any surplus tumour sample obtained at the time of acquired resistance to prior EGFR TKI
11. Men and women of childbearing potential must agree to use adequate contraception
12. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
13. Life expectancy greater or equal 12 weeks
14. Women of childbearing potential, including women who had their last menstrual period in the last 2 years, must have a negative serum or urine pregnancy test within 7 days before randomisation.
15. Patient is willing and able to comply with the protocol for the duration of the trial including undergoing treatment and scheduled visits and examinations including follow up.

Exclusion Criteria:

1. Prior systemic cytotoxic chemotherapy for advanced stage NSCLC Patients who had received previous adjuvant or neoadjuvant chemotherapy are eligible if the last dose of treatment was at least 12 months before randomisation.
2. Prior therapy with bevacizumab or other anti-angiogenic agent
3. Prior immune checkpoint inhibitor therapy
4. More than two lines of EGFR TKI therapy
5. Known small-cell lung carcinoma (SCLC) or high grade neuroendocrine carcinoma (if progression biopsy has been performed locally).
6. Squamous cell histologic subtype
7. Known EGFR T790M positive genotype by tissue on most recent EGFR TKI progression or ctDNA and have not received an approved EGFR TKI targeting T790M (e.g. a third-generation EGFR TKI such as osimertinib).
8. Active or untreated CNS metastases as determined by brain MRI

   - Patients with CNS metastases must be non-progressive by RECIST v1.1 and symptomatically stable with no ongoing requirement for corticosteroids as therapy for CNS disease; anticonvulsants at a stable dose allowed
9. Radiotherapy treatment to more than 30% of the bone marrow or with a wide field of radiation within 4 weeks of randomization.
10. Presence or history of a malignant disease that has been diagnosed and/or required therapy within the past 3 years. Exceptions to this exclusion include the following: completely resected basal cell and squamous cell skin cancers, and completely resected carcinoma in situ of any type.
11. Clear tumour infiltration into the thoracic great vessels (seen on imaging)
12. QTc of grade ≥3 according to CTCAE v5.0
13. Active autoimmune disease that has required systemic treatment in past 2 years. Patients with vitiligo, controlled type I diabetes mellitus on stable insulin, or residual autoimmune-related hypothyroidism only requiring hormone replacement or psoriasis not requiring systemic treatment are permitted
14. Active or uncontrolled HIV, tuberculosis, hepatitis B or C infection
15. Live attenuated vaccination within 4 weeks prior to randomisation.
16. Subject receiving any biologic drugs targeting the immune system (for example, TNF blockers, anakinra, rituximab, abatacept, or tocilizumab) within 6 weeks prior to treatment start.
17. History of idiopathic pulmonary fibrosis, organizing pneumonia, drug-induced pneumonitis, idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography scan. History of radiation pneumonitis in the radiation field (fibrosis) is permitted
18. Inadequately controlled hypertension (defined as systolic blood pressure >150 mmHg and/or diastolic blood pressure >100 mmHg)

    - Anti-hypertensive therapy to achieve these parameters is allowable.
19. Prior history of hypertensive crisis or hypertensive encephalopathy
20. Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent peripheral arterial thrombosis) within 6 months prior to randomization
21. History of haemoptysis (greater or equal 2.5mL of bright red blood per episode) within 1 month prior to randomization
22. Evidence of bleeding diathesis or coagulopathy (in the absence of therapeutic anticoagulation)
23. Current or recent (within 10 days before randomization) use of aspirin (>325 mg/day) or treatment with dipyramidole, ticlopidine, clopidogrel, and clostazol
24. Current use of full-dose oral or parenteral anticoagulants or thrombolytic agents for therapeutic purposes that has not been stable for >2 weeks prior to randomization

    * The use of full-dose oral or parenteral anticoagulants is permitted as long as the INR or aPTT is within therapeutic limits (according to the medical standard of the enrolling institution) and the patient has been on a stable dose of anticoagulants for at least 2 weeks prior to randomization.
    * Prophylactic anticoagulation for the patency of venous access devices is allowed, provided the activity of the agent results in an INR <1.5× ULN and aPTT is within normal limits within 14 days prior to randomization.
    * Prophylactic use of low-molecular-weight heparin (i.e., enoxaparin 40 mg/day) is permitted.
25. Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to the first dose of bevacizumab

    * Major surgery or significant traumatic injury 28 days prior to the first dose of bevacizumab.
    * Minor surgical procedure within 7 days, or placement of a vascular access device 2 days prior to the first dose of bevacizumab.
26. History of abdominal or tracheoesophageal fistula or gastrointestinal perforation within 6 months prior to randomization
27. Clinical signs of gastrointestinal obstruction or requirement for routine parenteral hydration, parenteral nutrition, or tube feeding
28. Evidence of abdominal free air not explained by paracentesis or recent surgical procedure
29. Serious, non-healing wound, active ulcer, or untreated bone fracture
30. Proteinuria, as demonstrated by urine dipstick or >1.0 g of protein in a 24-hour urine collection

    - All patients with greater or equal 2+ protein on dipstick urine analysis at baseline must undergo a 24 hour urine collection and must demonstrate lesser or equal 1 g of protein in 24 hours.
31. Any unresolved toxicities from prior therapy greater than CTCAE v5.0 grade 1 at the time of starting trial treatment with the exception of alopecia
32. History of hypersensitivity to the known active substances (atezolizumab, bevacizumab and chemotherapy drugs) or to any of the excipients.
33. History of hypersensitivity to Chinese Hamster Ovary (CHO) cell products or other recombinant human or humanised antibodies.
34. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements.
35. Women who are pregnant or in the period of lactation.
36. Sexually active men and women of childbearing potential who are not willing to use an effective contraceptive method during the trial and up to 6 months after discontinuing trial treatment
37. History of active diverticulitis

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2020-09-29 (Actual); Primary Completion 2024-07-22 (Actual); Study Completion 2024-07-22 (Actual)

PRIMARY OUTCOMES:
Progression-free survival (PFS) rate at 12 months according to RECIST v1.1 | 12 months from randomisation
  The primary objective of this study is to explore the clinical efficacy of atezolizumab and bevacizumab combined with chemotherapy in patients with EGFR-mutant advanced NSCLC after failure of standard EGFR TKIs.

SECONDARY OUTCOMES:
Adverse events according to CTCAE v5.0 | from the date of randomisation until 90 days after the last dose of protocol treatment
  To assess the safety and tolerability of the treatment.
Overall survival | through study completion, from the date of randomisation until death, including OS rate at 12 months.
  OS is defined as the time from the date of randomisation until death from any cause. Censoring will occur at the last follow-up date.
Objective response | From date of randomisation until date of treatment completion (until documented disease progression, death or any other causes), assessed up to 2 years.
  Objective response is defined as best overall response (CR or PR) across all assessment time-points according to RECIST v1.1, from randomisation until either the end of protocol treatment or the end of follow-up.
Quality of Life Core Questionnaire (EORTC QLQ-C30) | from baseline up to 12 months or until disease progression, whatever is first.
  Quality of life will be assessed by the European Organization for Research and Treatment of Cancer Quality of Life Core Questionnaire (EORTC QLQ-C30). The key QoL outcome is the time to deterioration (TTD) in the QLQ-C30 global health status/global QoL.
Quality of Life lung cancer-specific module (QLQ-LC13) | from baseline up to 12 months or until disease progression, whatever is first.
  Lung cancer associated symptoms will be measured by the lung cancer-specific module (QLQ-LC13).
Extra-cranial PFS | through study completion, from date of randomisation to documentation of PD outside the CNS, assessed up to 2 years
  Extra-cranial progression-free-survival is the time from randomisation to documentation of disease progression outside the central nervous system (CNS) as per RECIST v1.1 or death, whichever occurred first.
Intracranial PFS | through study completion, from date of randomisation to first documented radiographic evidence of CNS progression, assessed up to 2 years.
  Intracranial progression-free-survival is defined as the time from randomisation to first documented radiographic evidence of CNS progression. CNS progression is defined as progression due to newly developed CNS lesions and/or progression of pre-existing baseline CNS lesions.

CONTACTS AND LOCATIONS:
Locations (18):
- Germany (2):
  - LungenClinic Grosshansdorf, Großhansdorf
  - Asklepios Fachkliniken München-Gauting, München
- National University Hospital, Singapore, Singapore
- South Korea (2):
  - National Cancer Center, Goyang
  - Severance Hospital, Yonsei University Health System, Seoul
- Spain (10):
  - Hospital Teresa Herrera, A Coruña
  - ICO - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital De La Santa Creu I Sant Pau, Barcelona
  - Vall d'Hebron University Hospital, Barcelona
  - OSI Bilbao Basurto, Bilbao
  - Complejo Hospitalario de Jaén, Jaén
  - Hospital Universitario Insular Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Puerta de Hierro, Madrid
  - Hospital Universitario Fundacion Jimenez Díaz, Madrid
  - Hospital General de Valencia, Valencia
- Switzerland (3):
  - Hôpitaux Universitaires de Genève, Geneva
  - Kantonsspital St. Gallen, Sankt Gallen
  - UniversitätsSpital Zürich, Zurich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Soo RA, Vervita K, Fruh M, Cho BC, Majem M, Rodriguez Abreu D, Ribi K, Callejo A, Moran T, Domine Gomez M, Provencio M, Addeo A, Han JY, Ortega Granados AL, Reck M, Blasco A, Garcia Campelo R, Sala Gonzalez MA, Britschgi C, Roschitzki-Voser H, Ruepp B, Gasca-Ruchti A, Haberecker M, Dafni U, Peters S, Stahel RA; ETOP 15-19 ABC-lung collaborators. A randomised non-comparative phase II study of atezolizumab, bevacizumab and chemotherapy in EGFR-mutant NSCLC with acquired resistance - The ETOP 15-19 ABC-lung trial. Lung Cancer. 2025 Apr;202:108454. doi: 10.1016/j.lungcan.2025.108454. Epub 2025 Feb 20. PMID 40023017